CLINICAL TRIAL: NCT03404388
Title: Brain and Behavioral Influences on Motor Skill Learning in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Nora Fritz, Assistant Professor, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 122415M1E
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Masking Description: All participants will receive the same testing and training. A assessor blinded to whether the participant has received training will assess the Berg Balance Scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Balance Training
  Interventions: Behavioral: Balance Training

INTERVENTIONS:
Behavioral: Balance Training — 4 days of a challenging balance training task

SUMMARY:
Multiple Sclerosis (MS) is characterized by episodic attacks in which there are sharp declines in physical function. Although neurorehabilitation is the most promising clinical strategy for motor recovery in patients with MS, treatment responsiveness and outcomes are mixed. This is perhaps because each individual with MS has a different capacity to improve with rehabilitation, and this capacity may be based on a variety of baseline factors, such as disease duration, motivation, cognitive status and integrity of underlying brain structures. A better understanding of what "key ingredients" facilitate relearning of motor skills during neurorehabilitation is critically needed. Much of the focus of rehabilitation is on relearning motor skills. The initial stage of learning a motor skills often requires explicit concentration on the details of the movement. As one becomes more proficient in the motor skill, it becomes less attention-demanding and more automatic. Those who can perform motor skills more automatically will be better able to manage the additional demands of a secondary task; thus, capacity for dual-task performance can be used as an index of automaticity. Individuals with MS experience demyelination that impacts brain areas critical for motor learning. However, the specific clinical and pathological variables that facilitate capacity for motor learning in people with MS have not been identified. Identification of such variables could be leveraged to determine a patient's capacity to benefit from neurorehabilitation at the outset and potentially to maximize motor learning during rehabilitation for people with MS. Thus, there is an urgent need to determine the key ingredients most strongly associated with successful relearning of motor skills in MS patients.

Our long-term goal is to develop individualized rehabilitation for persons with MS. Our overall objective in this application is to identify clinical and pathological variables associated with successful relearning of motor skills. Our central hypothesis, based on preliminary data, is that the ability to learn to make new movements automatically occurs over a dynamic range and is a function of available cognitive processing speed and the integrity of corticospinal tract and superior cerebellar peduncles. We will test these hypotheses by recruiting 146 individuals with relapsing-remitting MS to participate in a mechanistic trial not designed to be a therapeutic intervention. Participants will complete baseline testing (including neuroimaging, cognitive testing and dual-task performance) followed by 4 consecutive days of training on a challenging balance task. After a 2-day washout period, participants will return for post-testing (including dual-task performance on a dual-balance and working memory task). The rationale for the proposed research is that identification of key ingredients associated with the capacity for motor skill acquisition would allow for more targeted rehabilitation programming, thereby improving patient outcomes and reducing health care expenses.

At the completion of the proposed research, we expect to understand more about the capacity for individuals with MS to improve with motor skill training, and some of the key ingredients that help predict successful shift toward task automaticity, one critical component of successful neurorehabilitation. The results of this proposal will facilitate the development of predictors of motor recovery, needed to improve rehabilitation outcomes for individuals with MS and other neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Relapsing-Remitting MS,
2. Patient Determined Disease Steps (PDDS) <6.5, indicating ability to ambulate with or without an assistive device (Hohol, 1999; Learmonth, 2013)
3. between the ages of 18 and 65;
4. stable medication regime for 3 months prior to enrollment, and
5. able to follow study-related commands.

Exclusion Criteria:

1. history of other neurological or neuromuscular conditions,
2. acute orthopedic conditions that prevent participation in the training,
3. steroid use <30 days prior to enrollment;
4. history of alcohol abuse;
5. presence of metallic implants, medical implants or exposure to metallic shrapnel incompatible with MRI,
6. pregnancy;
7. history of hospitalization for depression; and
8. depression as evidenced by a score of ≥10 on the Patient Health Questionnaire-9 (PHQ-9) (Kroenke, 2001), as depression has been shown to impact motor learning in persons with neurologic disorders (Subramanian, 2015).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Dual-Task Cost | Outcome will be assessed at baseline visit and post-test visit (1 week later)
  Performance of challenging balance task at the same time as a cognitive task

SECONDARY OUTCOMES:
Berg Balance Scale | Outcome will be assessed at baseline visit and post-test visit (1 week later)
  Clinical test of balance
Objective Balance Control | Outcome will be assessed at baseline visit and post-test visit (1 week later)
  Assessment of static and dynamic balance as well as anticipatory postural control with wearable sensors

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided